CLINICAL TRIAL: NCT03239340
Title: A Multicentre, Open-label, Single-arm, Molecular Profiling Study of Patients With EGFR Mutation-positive Locally Advanced or Metastatic NSCLC Treated With Osimertinib
Brief Title: A Molecular Profiling Study of Patients With EGFR Mutation-positive Locally Advanced or Metastatic NSCLC Treated With Osimertinib
Acronym: ELIOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5161C00003; 2017-002359-27 (EudraCT Number)
Record Dates: First submitted 2017-07-27; First posted 2017-08-04 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: EGFR Mutation Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Keywords: EGFR, NSCLC, Lung Cancer, Biopsy, Molecular Profiling
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental): An oral, potent, selective, irreversible inhibitor of both EGFR-tyrosine kinase inhibitor sensitizing and resistance mutations in non-small cell lung cancer
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib is an oral, potent, selective, irreversible inhibitor of both EGFR-tyrosine kinase inhibitor sensitizing and resistance mutations in non-small cell lung cancer with a significant selectivity margin over wild type EGFR.
  Other Names: TAGRISSO, AZD9291

SUMMARY:
A multicentre, open-label, single-arm, molecular profiling study of patients with EGFR mutation-positive locally advanced or metastatic NSCLC treated with osimertinib.

DETAILED DESCRIPTION:
Study design This is a phase II, open-label, single-arm tissue and plasma acquisition study assessing the efficacy, safety and underlying resistance mechanisms of osimertinib (80 mg orally, once daily) as first-line treatment in patients with locally advanced or metastatic EGFR mutation positive non-small cell lung cancer who are EGFR tyrosine kinase inhibitor treatment-naïve and eligible for first-line treatment. Participants with EGFR mutation-positive non-small cell lung cancer will be required to consent to 2 mandatory tumour biopsies to be considered for enrolment in this study. The first biopsy will be done prior to initiating treatment with osimertinib and the second biopsy will be obtained any time between Investigator assessed, Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1)-defined progression and before the start of any new anticancer treatment. A third optional biopsy may be taken during the course of treatment at the Investigator's discretion if the patient consents and if clinically feasible. Tumour tissue and plasma samples will be collected and examined for genetic and non genetic aberrations that may be important in determining response and resistance to the treatment that participants will receive as a part of their cancer care. Patients should continue on osimertinib until progression or until other treatment discontinuation criteria are met. However, if patients continue to show clinical benefit to treatment as judged by the Investigator, patients may continue to receive osimertinib beyond RECIST 1.1-defined progression. Therefore, there is no maximum duration of treatment. Tumour assessments will be performed at baseline and then every 8 weeks from study enrolment until 3.5 years, and then every 10 weeks until RECIST 1.1-defined. Patients will be followed up for a period of 28 days following discontinuation of osimertinib. Target patient population Male and female patients aged 18 years and over with locally advanced or metastatic pathologically confirmed adenocarcinoma of the lung, not amenable to curative surgery or radiotherapy. Patients will have a tumour that harbours one of the EGFR mutations known to be associated with EGFR tyrosine kinase inhibitor sensitivity, either alone or in combination with other EGFR mutations (EGFR mutation status determined by a local laboratory). Patients must be EGFR tyrosine kinase inhibitor treatment-naïve and eligible to receive first line treatment with osimertinib. Osimertinib is an oral, potent, selective, irreversible inhibitor of both EGFR tyrosine kinase inhibitor sensitizing and resistance mutations in non-small cell lung cancer with a significant selectivity margin over wild type EGFR. Osimertinib (80 mg orally, once daily) will be administered. Doses may be reduced to 40 mg if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior
2. Patients aged 18 years or older
3. Patients with histological confirmation of locally advanced or metastatic NSCLC
4. Patients with M1 stage according to the Tumor, Node and Metastasis Classification of Malignant Tumours (TNM)
5. Patients with an EGFR deletion or mutation known (from tumour biopsy or plasma) to be associated with EGFR TKI sensitivity
6. Existence of measurable or evaluable disease (as per RECIST 1.1 criteria).
7. Possibility of obtaining sufficient tissue sample, via a biopsy or surgical resection of the primary tumour or metastatic tumour tissue
8. WHO performance status 0-1
9. Life expectancy ≥12 weeks
10. Capacity to swallow
11. Patients able to complete study and within geographical proximity allowing for adequate follow up
12. Resolution of all acute toxic effects of previous anticancer therapy
13. Female patients must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of childbearing potential
14. Male patients must be willing to use barrier contraception

Exclusion Criteria:

1. Locally advanced lung cancer candidate for curative treatment through radical surgery and/or radio(chemo)therapy
2. Patients diagnosed with another lung cancer subtype
3. Patients with an EGFR exon 20 insertion
4. Patients with just one measurable or evaluable tumour lesion that has been resected or irradiated prior to their enrolment in the study
5. Second active neoplasia
6. Treatment with an investigational drug within five half-lives of the compound
7. Participation in another clinical study with an investigational product (IP) during the last 3 weeks before the first day of study treatment
8. Patients who have received prior immunotherapies
9. Patients who have received prior EGFR treatments for lung cancer
10. Patients who have received prior treatment with an EGFR TKI including in the adjuvant setting
11. Patients who have received previous treatment for metastatic or stage IV disease
12. Prior treatment with cytotoxic chemotherapy for advanced NSCLC
13. Patients with a history of cancer that has been completely treated, with no evidence of malignant disease currently cannot be enrolled in the study if their chemotherapy was completed less than 6 months prior and/or have received a bone marrow transplant less than 2 years before the first day of study treatment
14. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy
15. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses or active infection (eg, patients receiving treatment for infection) including hepatitis C and human immunodeficiency virus (HIV), or active uncontrolled Hepatitis B virus (HBV) infection.
16. Patients who have had a surgical procedure unrelated to the study within 14 days or major surgery within 1 month prior to the administration of the study drug
17. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis
18. Any of the following cardiac criteria: Mean resting QT interval corrected for heart rate (QTc) more than 470 msec, obtained from 3 ECGs, using the screening clinic ECG machine derived QTc value. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, hypomagnesaemia, hypocalcaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
19. Spinal cord compression, symptomatic and unstable brain metastases except for those patients who have completed definitive therapy, and have had a stable neurological status for at least 2 weeks after completion of definitive therapy. 20.Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib

21.Inadequate bone marrow reserve or organ function 22.Female patients who are breastfeeding 23.Patients currently receiving medications or herbal supplements known to be potent inducers of cytochrome (CYP) 3A4.

24.Patient unwilling to undergo a biopsy at the time of disease progression 25.History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib 26.Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements 27.Involvement in the planning and/or conduct of the study 28.Previous enrolment in the present study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zosia Piotrowska, MD, Principal Investigator — Massachusetts General Hospital
Locations (23):
- United States (3):
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
- Italy (6):
  - Research Site, Brescia
  - Research Site, Meldola
  - Research Site, Monza
  - Research Site, Parma
  - Research Site, Roma
  - Research Site, Terni
- Malaysia (5):
  - Research Site, Johor Bahru
  - Research Site, Kuantan
  - Research Site, Kuching
  - Research Site, Lembah Pantai
  - Research Site, Pulau Pinang
- South Korea (4):
  - Research Site, Busan
  - Research Site, Cheongiu
  - Research Site, Seongnam
  - Research Site, Seoul
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00003&attachmentIdentifier=0512bdf7-7e91-4862-b078-e8c798059269&fileName=235434_CSR_Synopsis_28-June-24_Redacted_Approved_PDF_A.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00003&attachmentIdentifier=38f2807f-f212-4590-8e86-5b2d13cb3772&fileName=235434_Protocol_13Aug_24_Redacted_Approved_PDF_A.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00003&attachmentIdentifier=806e2b73-bfa4-4a78-890a-f0655e38acb4&fileName=235434_SAP_13Aug_24_Redacted_Approved_PDF_A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 30 May 2018 (First subject in) and analyses presented in this results form are based on a final data cut-off of 18 July 2023 and final database lock of 15 December 2023.
Pre-assignment Details: Participants meeting eligibility criteria predefined in protocol were enrolled in the study. All the assessments were performed as per the schedule of the assessments.
Groups:
- Osimertinib 80mg: Participants received Osimertinib 80mg orally once daily.
Period: Overall Study
Arm/Group | Osimertinib 80mg
Started | 154
Completed | 33
Not Completed | 121
Not completed — Other | 26
Not completed — Patients who are ongoing in the study at DCO | 10
Not completed — Death | 40
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 16
Not completed — Withdrawal by Subject | 27

BASELINE CHARACTERISTICS:
Arm/Group | Osimertinib 80mg
Number analyzed (Participants) | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 62
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 30
  Black or African American | 5
  Asian | 118
  Other | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic | 6
  Not Hispanic or Latino | 148

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Given Tumour Genetic and Proteomic Marker at the Point of Disease Progression
Description: The frequency of genetic and proteomic markers at disease progression regardless of their prevalence was evaluated.
Time Frame: Genetic and proteomic markers were assessed at baseline and progression (up to 5 years after baseline)
Population: The primary analysis set included all patients with evaluable paired biopsies, which were defined as follows: the first biopsy was taken prior to osimertinib treatment, and the second biopsy was taken at any time between Investigator-assessed RECIST 1.1-defined progression and before the start of any new anticancer treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Osimertinib 80 mg: Participants received Osimertinib 80mg orally once daily.
Arm/Group | Osimertinib 80 mg
Number analyzed (Participants) | 51
Percentage of participants
  AKT2; Copy Number Alteration: Type; amplification | 2.0 [0.05 to 10.45]
  ALK; Rearrangement | 3.9 [0.48 to 13.46]
  APC; Copy Number Alteration; Type: loss | 2.0 [0.05 to 10.45]
  ARAF; Copy Number Alteration; Type: amplification | 3.9 [0.48 to 13.46]
  ASXL1; Short Variant; Type: Q588* | 2.0 [0.05 to 10.45]
  ATRX; Short Variant; Type: P599fs*22 | 2.0 [0.05 to 10.45]
  AXL; Copy Number Alteration; Type: amplification | 2.0 [0.05 to 10.45]
  BCL2L2; Copy Number Alteration; Type: amplification | 3.9 [0.48 to 13.46]
  BRAF; Rearrangement | 2.0 [0.05 to 10.45]
  BRAF; Short variant; Type: G469A | 2.0 [0.05 to 10.45]
  BRAF; Short variant Type: V600E | 3.9 [0.48 to 13.46]
  CBL; Short Variant; Type: R149Q | 2.0 [0.05 to 10.45]
  CCND1 Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  CCNE1 Copy Number Alteration Type: amplification | 5.9 [1.23 to 16.24]
  CDK4 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  CDK6 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  CDKN1B Short Variant Type: S2* | 2.0 [0.05 to 10.45]
  CDKN2A Copy Number Alteration Type: loss | 15.7 [7.02 to 28.59]
  CDKN2A; Short Variant Type: P38L | 2.0 [0.05 to 10.45]
  CDKN2B Copy Number Alteration Type: loss | 15.7 [7.02 to 28.59]
  CRKL Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  CUL4A Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  DIS3 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  EGFR Copy Number Alteration Type: amplification | 11.8 [4.44 to 23.87]
  EGFR Rearrangement | 2.0 [0.05 to 10.45]
  EGFR Short Variant Type: C797S | 7 [5.70 to 26.26]
  EGFR Short Variant Type: L858R | 2.0 [0.05 to 10.45]
  EMSY Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  ERBB2 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  FANCG Rearrangement | 2.0 [0.05 to 10.45]
  FGF10 Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  FGF14; Copy Number Alteration; Type: amplification | 2.0 [0.05 to 10.45]
  FGF19 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  FGFR1 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  FGFR3 Rearrangement | 2.0 [0.05 to 10.45]
  FGFR4 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  HGF Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  HRAS Short Variant Type: Q61R | 2.0 [0.05 to 10.45]
  IDH1 Short Variant Type: R132L | 2.0 [0.05 to 10.45]
  IGF1R Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  IRS2 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  KRAS Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  LYN Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  MAP2K1 Short Variant Type: E102_I103del | 2.0 [0.05 to 10.45]
  MCL1 Copy Number Alteration Type: amplification | 5.9 [1.23 to 16.24]
  MDM2 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  MET Copy Number Alteration Type: amplification | 17.6 [8.40 to 30.87]
  MTAP Copy Number Alteration Type: loss | 13.7 [5.70 to 26.26]
  MYC Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  MYCN Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  NF1 Short Variant Type: M1I | 2.0 [0.05 to 10.45]
  NFE2L2 Short Variant Type: D29N | 2.0 [0.05 to 10.45]
  NFKBIA Copy Number Alteration Type: amplification | 9.8 [3.26 to 21.41]
  NKX2-1 Copy Number Alteration Type: amplification | 9.8 [3.26 to 21.41]
  NOTCH3 Rearrangement | 2.0 [0.05 to 10.45]
  NTRK1 Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  PARP1 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  PDGFRB Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  PIK3CA Short Variant Type: E542K | 2.0 [0.05 to 10.45]
  PIM1 Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  RAD21 Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  RB1 Copy Number Alteration Type: loss | 3.9 [0.48 to 13.46]
  RB1 Short Variant Type: Q846* | 2.0 [0.05 to 10.45]
  RICTOR Copy Number Alteration Type: amplification | 7.8 [2.18 to 18.88]
  SMAD4 Rearrangement | 2.0 [0.05 to 10.45]
  SMAD4 Short Variant Type: W524L | 2.0 [0.05 to 10.45]
  SPEN Short Variant Type: D2047fs*17 | 2.0 [0.05 to 10.45]
  STK11 Copy Number Alteration Type: loss | 2.0 [0.05 to 10.45]
  STK11 Short Variant Type: K269fs*18 | 2.0 [0.05 to 10.45]
  TERC Copy Number Alteration Type: amplification | 2.0 [0.05 to 10.45]
  TERT Short Variant Type: promoter -146C>T | 2.0 [0.05 to 10.45]
  TET2 Short Variant Type: Q916* | 2.0 [0.05 to 10.45]
  TET2 Short Variant Type: V1862fs*13 | 2.0 [0.05 to 10.45]
  TP53 Short Variant Type: R213* | 2.0 [0.05 to 10.45]
  WHSC1L1 Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]
  ZNF703 Copy Number Alteration Type: amplification | 3.9 [0.48 to 13.46]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose of osimertinib until the date of Investigator assessed Response Evaluation Criteria in Solid Tumours (RECIST) 1.1-defined progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anticancer therapy prior to progression.
Time Frame: From date of first dose until date of progression or death (by any cause in the absence of recurrence), up to 5 years
Population: The full analysis set included all patients who received at least one dose of Osimertinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib 80 mg
Number analyzed (Participants) | 154
Months | 16.4 [12.7 to 20.3]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the number (%) of patients with at least one visit response of complete response (CR) or partial response (PR) that is confirmed at least 4 weeks later.
Time Frame: From date of first dose until progression, or last evaluable assessment in the absence of progression, up to 5 years
Population: The full analysis set included all patients who received at least one dose of Osimertinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Osimertinib 80 mg
Number analyzed (Participants) | 154
Percentage of participants | 73.4 [65.66 to 80.17]

4. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time from the date of first documented response, (that is subsequently confirmed) until date of documented progression or death in the absence of disease progression, the end of response should coincide with the date of progression or death from any cause used for the PFS endpoint. The time of the initial response will be defined as the latest of the dates contributing towards the first visit that was CR or PR that was subsequently confirmed.
Time Frame: From date of first documentation of complete/partial response until the date of progression, or last evaluable RECIST assessment for participants that did not progress within 2 missed visits of last assessment, up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib. The Duration of response is calculated for only participants with a confirmed response. Participants must have had measurable disease at baseline to be included in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib 80 mg
Number analyzed (Participants) | 113
Months | 18.8 [14.2 to 22.3]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as percentage of patients with confirmed complete response, confirmed partial response or with stable disease.
Time Frame: 8 weeks
Population: The full analysis set included all patients who received at least 1 dose of osimertinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Osimertinib 80 mg
Number analyzed (Participants) | 154
Percentage of participants | 94.8 [90.02 to 97.73]

6. Secondary Outcome: Time to Treatment Discontinuation or Death (TTD)
Description: TTD is defined as the time from the date of first dose of osimertinib to the earliest of treatment discontinuation or death.
Time Frame: From date of first dose to treatment discontinuation or death (by any cause in the absence of recurrence), up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Osimertinib 80 mg: Participants received Osimertinib 80 mg orally once daily with epidermal growth factor receptor (EGFR).
Arm/Group | Osimertinib 80 mg
Number analyzed (Participants) | 154
Months | 20.0 [16.3 to 23.8]

7. Secondary Outcome: Time to First Subsequent Therapy or Death (TFST)
Description: TFST is defined as the time from the date of first dose of osimertinib to the earlier of the date of anticancer therapy start date following study treatment discontinuation, or death.
Time Frame: From date of first dose to start of subsequent anticancer therapy or death (by any cause in the absence of recurrence), up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Osimertinib 80 mg: Participants received Osimertinib 80 mg orally once daily.
Arm/Group | Osimertinib 80 mg
Number analyzed (Participants) | 154
Months | 32.1 [24.0 to 47.7]

8. Secondary Outcome: PFS in Patient Subgroups Defined by Molecular Profile: Epidermal Growth Factor Receptor (EGFR) Tumor Mutation at Baseline
Description: PFS is defined as the time from first dose of osimertinib until the date of Investigator assessed Response Evaluation Criteria in Solid Tumours (RECIST) 1.1-defined progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anticancer therapy prior to progression. PFS was analysed in patient subgroups defined by molecular profile, including but not limited to: EGFR tumor mutation at baseline-Exon19del or L858R
Time Frame: From date of first dose until date of progression or death (by any cause in the absence of recurrence), up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Exon19del: Participants with Exon19del received Osimertinib 80mg orally once daily.
- L858R: Patient with L858R received Osimertinib 80 mg orally one daily.
Arm/Group | Exon19del | L858R
Number analyzed (Participants) | 85 | 58
Months | 22.0 [16.0 to 27.6] | 12.9 [10.8 to 18.2]

9. Secondary Outcome: PFS in Patient Subgroups Defined by Molecular Profile: Detectable in Plasma-Derived ctDNA at Baseline
Description: PFS is defined as the time from first dose of osimertinib until the date of Investigator assessed Response Evaluation Criteria in Solid Tumours (RECIST) 1.1-defined progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anticancer therapy prior to progression. PFS was analysed in patient subgroups defined by molecular profile, including but not limited to: Exon19del or L858R detectable in plasma derived circulating tumour deoxyribonucleic acid (ctDNA) at baseline.
Time Frame: From date of first dose until date of progression or death (by any cause in the absence of recurrence), up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Exon19del | L858R
Number analyzed (Participants) | 62 | 46
Months | 19.6 [12.7 to 24.0] | 13.7 [9.0 to 18.2]

10. Secondary Outcome: ORR in Patient Subgroups Defined by Molecular Profile: EGFR Tumor Mutation at Baseline
Description: ORR is defined as the number (%) of patients with at least one visit response of complete response or partial response that is confirmed at least 4 weeks later. ORR was analysed in patient subgroups defined by molecular profile: EGFR tumor mutation at baseline-Exon19del or L858R
Time Frame: From date of first dose until progression, or last evaluable assessment in the absence of progression, up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- L858R: Participants with L858R received Osimertinib 80mg orally once daily.
Arm/Group | Exon19del | L858R
Number analyzed (Participants) | 85 | 58
Percentage of participants | 82.4 [72.57 to 89.77] | 69.0 [55.46 to 80.46]

11. Secondary Outcome: ORR in Patient Subgroups Defined by Molecular Profile: Detectable in Plasma Derived ctDNA at Baseline
Description: ORR is defined as the number (%) of patients with at least one visit response of complete response or partial response that is confirmed at least 4 weeks later. ORR was analysed in patient subgroups defined by molecular profile: Exon19del or L858R detectable in plasma derived ctDNA at baseline.
Time Frame: From date of first dose until progression, or last evaluable assessment in the absence of progression, up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Exon19del | L858R
Number analyzed (Participants) | 62 | 46
Percentage of participants | 85.5 [74.22 to 93.14] | 71.7 [56.54 to 84.01]

12. Secondary Outcome: TTD in Patient Subgroups Defined by Molecular Profile: EGFR Tumor Mutation at Baseline
Description: TTD is defined as the time from the date of first dose of osimertinib to the earliest of treatment discontinuation or death. TTD was analysed in patient subgroups defined by molecular profile: EGFR tumor mutation at baseline-Exon19del or L858R
Time Frame: as for outcome 6
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Exon19del 80 mg: Participants with Exon19del received Osimertinib 80mg orally once daily.
Arm/Group | Exon19del 80 mg | L858R
Number analyzed (Participants) | 85 | 58
Months | 25.5 [19.6 to 32.1] | 16.5 [12.1 to 21.7]

13. Secondary Outcome: TTD in Patient Subgroups Defined by Molecular Profile: Detectable in Plasma Derived ctDNA at Baseline
Description: TTD is defined as the time from the date of first dose of osimertinib to the earliest of treatment discontinuation or death. TTD was analysed in patient subgroups defined by molecular profile: Exon19del or L858R detectable in plasma derived ctDNA at baseline.
Time Frame: as for outcome 6
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Exon19del 80 mg | L858R
Number analyzed (Participants) | 62 | 46
Months | 24.5 [17.8 to 29.6] | 16.5 [12.1 to 21.4]

14. Secondary Outcome: Tumour Shrinkage/Depth of Response in Patient Subgroups Defined by Molecular Profile: EGFR Tumor Mutation at Baseline
Description: Tumour shrinkage is defined as the best change from baseline in the sum of diameters of target lesions, in patient subgroups defined by molecular profile: EGFR tumor mutation at baseline-Exon19del or L858R. A negative change denotes a reduction in target lesion size.
Time Frame: From date of first dose until last recorded post baseline RECIST target lesion assessment scan, up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Exon19del | L858R
Number analyzed (Participants) | 83 | 55
Percentage change | -59.68 [-100.0 to 6.5] | -54.29 [-100.0 to 7.6]

15. Secondary Outcome: Tumour Shrinkage/Depth of Response in Patient Subgroups Defined by Molecular Profile: Detectable in Plasma Derived ctDNA at Baseline
Description: Tumour shrinkage is defined as the best change from baseline in the sum of diameters of target lesions, in patient subgroups defined by molecular profile: Exon19del or L858R detectable in plasma derived ctDNA at baseline. A negative change denotes a reduction in target lesion size.
Time Frame: From date of first dose until last recorded post baseline RECIST target lesion assessment scan, up to 5 years
Population: The full analysis set included all patients who received at least 1 dose of Osimertinib.
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Exon19del | L858R
Number analyzed (Participants) | 60 | 44
Percentage change | -60.80 [-100.0 to 6.5] | -58.33 [-100.0 to 7.6]

ADVERSE EVENTS:
Time Frame: From Day 1 to Follow-up (28 days post last dose) up to 5 years
Arm/Group | Osimertinib 80 mg
All-Cause Mortality (participants affected / at risk) | 40/154
Serious Adverse Events (participants affected / at risk) | 53/154
Other Adverse Events (participants affected / at risk) | 148/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib 80 mg (N=154)
COVID-19 (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 12
Pneumonia aspiration (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Confusional state (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Asthenia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Platelet count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib 80 mg (N=154)
COVID-19 (Infections and infestations) | 14
Paronychia (Infections and infestations) | 36
Upper respiratory tract infection (Infections and infestations) | 24
Urinary tract infection (Infections and infestations) | 16
Anaemia (Blood and lymphatic system disorders) | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 27
Insomnia (Psychiatric disorders) | 10
Dizziness (Nervous system disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 32
Headache (Nervous system disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 63
Gastritis (Gastrointestinal disorders) | 8
Mouth ulceration (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 17
Stomatitis (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 14
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 21
Dry skin (Skin and subcutaneous tissue disorders) | 30
Pruritus (Skin and subcutaneous tissue disorders) | 23
Rash (Skin and subcutaneous tissue disorders) | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Asthenia (General disorders) | 13
Fatigue (General disorders) | 11
Alanine aminotransferase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 14
Gamma-glutamyltransferase increased (Investigations) | 9
Platelet count decreased (Investigations) | 11
Weight decreased (Investigations) | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03239340/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT03239340/SAP_001.pdf